CLINICAL TRIAL: NCT02452476
Title: A DOUBLE BLIND, RANDOMIZED, CONTROLLED STUDY TO INVESTIGATE THE EFFICACY AND SAFETY OF SYNTHETIC SURFACTANT (CHF 5633) IN COMPARISON TO PORCINE SURFACTANT (PORACTANT ALFA, CUROSURF®) IN THE TREATMENT OF PRETERM NEONATES WITH RESPIRATORY DISTRESS SYNDROME
Brief Title: A Double Blind, Randomized, Controlled Study to Evaluate CHF 5633 (Synthetic Surfactant) and Poractant Alfa in Neonates With Respiratory Distress Syndrome (RDS) (POC)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chiesi Farmaceutici S.p.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CCD-05633AA1-02
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Results first posted 2021-06-23 (Actual); Last update posted 2021-08-13 (Actual); Status verified 2021-07

CONDITIONS: Respiratory Distress Syndrome, Newborn
Keywords: neonates, pulmonary surfactant
MeSH Terms: conditions — Respiratory Distress Syndrome, Newborn | interventions — CHF5633; poractant alfa

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- CHF5633 (Experimental): Single dose within 24 hours from birth
  Interventions: Drug: CHF5633
- Poractant alfa (Active Comparator): Single dose within 24 hours from birth
  Interventions: Drug: Poractant alfa

INTERVENTIONS:
Drug: CHF5633 — Rescue treatment (if needed)
  Arms: CHF5633
Drug: Poractant alfa — Rescue treatment (if needed)
  Arms: Poractant alfa

SUMMARY:
A multicenter, double blind, randomized, single dose, active-controlled study to investigate the efficacy and safety of synthetic surfactant (CHF 5633) in comparison to porcine surfactant (Poractant alfa, Curosurf ®) in the treatment of preterm neonates with respiratory distress syndrome. Main objectives of this study are to investigate the short term efficacy profile of CHF 5633 vs. porcine surfactant (Poractant Alfa, Curosurf®) in terms of reduced oxygen requirement and ventilatory support and to evaluate the mid-term efficacy profile in terms of reduced incidence of bronchopulmonary dysplasia (BPD) and mortality/BPD rate at 36 weeks post menstrual age (PMA), mortality rate at 28 days and 36 weeks PMA, RDS-associated mortality through 14 days of age and other major co-morbidities of prematurity.

Inclusion criteria are: Written parental informed consent, inborn preterm neonates of either sex with a gestational age of 24+0 weeks up to 29+6 weeks, clinical course consistent with RDS, requirement of endotracheal surfactant administration within 24 hours from birth, fraction of inspired oxygen (FiO2) ≥0.30 for babies 24+0 to 26+6 weeks and FiO2 ≥0.35 for babies 27+0 to 29+6 weeks to maintain arterial oxygen saturation by pulse oximetry (SpO2) between 88-95%.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained by parents/legal representative (according to local regulation) prior to any study-related procedures
2. Inborn preterm neonates of either sex with a gestational age of 24+0 weeks up to 29+6 weeks
3. Clinical course consistent with RDS
4. Requirement of endotracheal surfactant administration within 24 hours from birth
5. Fraction of inspired oxygen (FiO2) ≥0.30 for babies 24+0 to 26+6 weeks and FiO2 ≥0.35 for babies 27+0 to 29+6 weeks to maintain SpO2 between 88-95%

Exclusion Criteria:

1. Use of surfactant prior to study entry and need for intratracheal administration of any other treatment (e.g. nitric oxide)
2. Known genetic or chromosomal disorders, major congenital anomalies (cardiac malformations, myelomeningocele etc)
3. Maternal drug abuse (heroin, methadone, methamphetamine, or cocaine) or significant alcohol consumption during pregnancy
4. Mothers with prolonged rupture of the membranes (>21 days duration)
5. Strong suspicion of congenital pneumonia/infection, sepsis
6. Presence of air leaks prior to study entry
7. Evidence of severe birth asphyxia
8. Neonatal seizures prior to study entry
9. Any condition that, in the opinion of the Investigator, would place the neonate at undue risk
10. Participation in another clinical trial of any placebo, drug or biological substance conducted under the provisions of a protocol.

Ages: 1 Hour to 24 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 123 (Actual)
Dates: Start 2016-01-21 (Actual); Primary Completion 2018-05-24 (Actual); Study Completion 2018-05-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rangasamy Ramanathan, MD, Principal Investigator — Division of Neonatology, Department of Pediatrics, LAC+USC Medical Center and Good Samaritan Hospital, Keck School of Medicine of USC, Los Angeles, CA, USA
Locations (23):
- United States (23):
  - University of South Alabama - USA Children's and Women's Hospital, Mobile, Alabama
  - LAC + USC Medical Center, Keck School of Medicine, Los Angeles, California
  - UC Irvine Medical Center, Orange, California
  - Sharp Mary Birch Hospital, San Diego, California
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Plantation General Hospital (Sheridan Clinical Research, Inc.), Plantation, Florida
  - Jatinder Bhatia, Augusta, Georgia
  - Indiana University School of Medicine, Indianapolis, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - University of Louisville Research Foundation, Inc., Louisville, Kentucky
  - Floating Hospital for Children at Tufts Medical Center, Boston, Massachusetts
  - Baystate Children's Hospital / Baystate Medical Center, Springfield, Massachusetts
  - Winthrop University Hospital, Mineola, New York
  - Kings County Hospital Center, New York, New York
  - Sergio G. Golombek, Valhalla, New York
  - Martha Naylor, Greenville, North Carolina
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Krishnamurthy Sekar, Oklahoma City, Oklahoma
  - Hahnemann University Hospital, Philadelphia, Pennsylvania
  - Texas Tech University Health Sciences Center, El Paso, Texas
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
  - West Virginia University, Morgantown, West Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ramanathan R, Biniwale M, Sekar K, Hanna N, Golombek S, Bhatia J, Naylor M, Fabbri L, Varoli G, Santoro D, Del Buono D, Piccinno A, Dammann CE. Synthetic Surfactant CHF5633 Compared with Poractant Alfa in the Treatment of Neonatal Respiratory Distress Syndrome: A Multicenter, Double-Blind, Randomized, Controlled Clinical Trial. J Pediatr. 2020 Oct;225:90-96.e1. doi: 10.1016/j.jpeds.2020.06.024. Epub 2020 Jun 14. PMID 32553868

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CHF5633 | Poractant Alfa
Started | 64 | 59
Completed | 53 | 49
Not Completed | 11 | 10
Not completed — Death | 4 | 7
Not completed — Lost to Follow-up | 1 | 1
Not completed — Physician Decision | 1 | 1
Not completed — Not treated | 5 | 1

BASELINE CHARACTERISTICS:
Population: Premature infants were screened according to study inclusion and exclusion criteria. Overall, 123 patients were randomized (6 patients were withdrawn before treatment start).
  Overall, 117 patients received double-blind treatment. The baseline characteristics shown in the table below are based on the intention-to-treat (ITT) population (ITT=All randomized patients who received at least one dose of study medication and with at least one available evaluation of efficacy after the baseline).
Groups:
- Total: Total of all reporting groups
Arm/Group | CHF5633 | Poractant Alfa | Total
Number analyzed (Participants) | 56 | 57 | 113
Age, Continuous [Mean (Standard Deviation); unit: hours] | 1.87 (4.12) | 1.26 (3.21) | 1.56 (3.69)
Age, Continuous [Mean (Standard Deviation); unit: weeks] — Gestational age.
  weeks | 27.01 (1.79) | 26.72 (1.90) | 26.86 (1.84)
Age, Customized [Count of Participants; unit: Participants] — Gestational age group
  Participants
    24 to 26 Weeks | 26 | 32 | 58
    27 to 29 Weeks | 30 | 25 | 55
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 29 | 61
  Male | 24 | 28 | 52
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 15 | 17 | 32
  Not Hispanic or Latino | 37 | 34 | 71
  Unknown or Not Reported | 4 | 6 | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 1
  Black or African American | 23 | 19 | 42
  White | 25 | 26 | 51
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 7 | 8 | 15
Region of Enrollment [Number; unit: participants]
  United States | 56 | 57 | 113
APGAR Score [Mean (Standard Deviation); unit: units on a scale] — APGAR Score at birth to summarize the health of a newborn.The Apgar score is based on a total score of 1 to 10. The higher the score, the better the baby is doing after birth. A score of 7, 8, or 9 is normal and is a sign that the newborn is in good health.
  units on a scale | 6.3 (1.8) | 5.9 (1.9) | 6.1 (1.9)
Birth weight [Mean (Standard Deviation); unit: gram] | 862.0 (247.2) | 903.6 (310.2) | 883.0 (280.3)

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Requirement and Ventilatory Support -- SpO2/FiO2 Ratio
Description: SpO2/FiO2 ratio
  The oxygen requirement and ventilatory support were assessed through arterial oxygen saturation, measured by pulse oximetry (SpO2 [%]) and ventilator settings, by measuring fraction of inspired oxygen (FiO2[%]) and SpO2/FiO2. Results are shown as change from baseline, summarized at post-treatment timepoints.
  Definitions:
  SpO2=Arterial Oxygen saturation by pulse oximetry; FiO2=Fraction of inspired oxygen; Baseline=The last pre-dose measurement taken on Day -1.
Time Frame: Post-treatment Day 1: 30 min, at 1h, 3h, 6h, 12h, 18h, 24 h; Day 2, 3, 5, and 7
Population: Intention-to-Treat Population (ITT). All randomized patients who received at least one dose of study medication and with at least one available evaluation of efficacy after the baseline.
Measure: Least Squares Mean (95% Confidence Interval); unit: SpO2/FiO2 ratio
Arm/Group | CHF5633 | Poractant Alfa
Number analyzed (Participants) | 56 | 57
SpO2/FiO2 ratio
  Day 1, 30 min | 3.33 [3.02 to 3.63] | 3.31 [3.00 to 3.61]
  Day 1, 1 h | 3.36 [3.07 to 3.66] | 3.55 [3.26 to 3.84]
  Day 1, 3 h | 3.58 [3.33 to 3.83] | 3.68 [3.44 to 3.93]
  Day 1, 6 h | 3.77 [3.52 to 4.02] | 3.87 [3.63 to 4.12]
  Day 1, 12 h | 3.89 [3.65 to 4.13] | 3.78 [3.54 to 4.01]
  Day 1, 18 h | 3.82 [3.59 to 4.04] | 3.74 [3.52 to 3.97]
  Day 1, 24 h | 3.72 [3.47 to 3.98] | 3.64 [3.38 to 3.89]
  Day 2: number analyzed (Participants) | 56 | 53
  Day 2 | 3.61 [3.35 to 3.86] | 3.63 [3.38 to 3.88]
  Day 3: number analyzed (Participants) | 54 | 53
  Day 3 | 3.75 [3.48 to 4.01] | 3.78 [3.52 to 4.05]
  Day 5: number analyzed (Participants) | 54 | 50
  Day 5 | 3.83 [3.56 to 4.10] | 3.88 [3.61 to 4.15]
  Day 7: number analyzed (Participants) | 53 | 51
  Day 7 | 3.74 [3.47 to 4.00] | 3.73 [3.46 to 3.99]
Statistical Analysis 1: Comparison: CHF5633 vs Poractant Alfa; Day 1, 30 min post dose. SpO2/FiO2 and FiO2 (%) over the first 24 hours: analyzed using a linear mixed model for repeated measures (MMRM) including treatment, timepoint, treatment by timepoint interaction, investigational site and gestational age (GA) group as fixed effects, and predose values as covariates. The adjusted mean difference between treatments, and their 95% confidence intervals (CIs) at each timepoint and averaged over the first 24 hours were estimated by the model; Test type: Superiority; p = 0.930, Mixed model for repeated measurements; Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.40 to 0.44]
Statistical Analysis 2: Comparison: CHF5633 vs Poractant Alfa; Day 1, 1 h post dose; Test type: Superiority; p = 0.346, Mixed model for repeated measurements; Mean Difference (Final Values) = -0.19, 95% CI 2-sided [-0.59 to 0.21]
Statistical Analysis 3: Comparison: CHF5633 vs Poractant Alfa; Day 1, 3 h post dose; Test type: Superiority; p = 0.549, Mixed model for repeated measurements; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.43 to 0.23]
Statistical Analysis 4: Comparison: CHF5633; Day 1, 6 h post dose; Test type: Superiority; p = 0.539, Mixed model for repeated measurements; Mean Difference (Final Values) = -0.10, 95% CI 2-sided [-0.43 to 0.23]
Statistical Analysis 5: Comparison: CHF5633 vs Poractant Alfa; Day 1, 12 h post dose; Test type: Superiority; p = 0.491, Mixed model for repeated measurements; Mean Difference (Final Values) = 0.11, 95% CI 2-sided [-0.21 to 0.43]
Statistical Analysis 6: Comparison: CHF5633 vs Poractant Alfa; Day 1, 18 h post dose; Test type: Superiority; p = 0.623, Mixed model for repeated measurements; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.22 to 0.37]
Statistical Analysis 7: Comparison: CHF5633 vs Poractant Alfa; Day 1, 24 h post dose; Test type: Superiority; p = 0.608, Mixed model for repeated measurements; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-0.25 to 0.43]
Statistical Analysis 8: Comparison: CHF5633 vs Poractant Alfa; Day 2, post dose SpO2/FiO2 was compared between treatments at the remaining post-treatment time points (i.e., Days 2, 3, 5, 7): analyzed using mixed model including treatment, investigational site and gestational age group as fixed effects and pre-dose ratio as covariate; Test type: Superiority; p = 0.869, Mixed Models Analysis; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.35 to 0.30]
Statistical Analysis 9: Comparison: CHF5633 vs Poractant Alfa; Day 3, post dose; Test type: Superiority; p = 0.833, Mixed Models Analysis; Mean Difference (Final Values) = -0.04, 95% CI 2-sided [-0.38 to 0.31]
Statistical Analysis 10: Comparison: CHF5633 vs Poractant Alfa; Day 5, post dose; Test type: Superiority; p = 0.772, Mixed Models Analysis; Mean Difference (Final Values) = -0.05, 95% CI 2-sided [-0.39 to 0.29]
Statistical Analysis 11: Comparison: CHF5633 vs Poractant Alfa; Day 7, post dose; Test type: Superiority; p = 0.963, Mixed Models Analysis; Mean Difference (Final Values) = 0.01, 95% CI 2-sided [-0.33 to 0.35]

2. Primary Outcome: Fraction of Inspired Oxygen (FiO2) (Percent) During the First 24 h and up to Day 7
Description: Fraction of inspired oxygen (FiO2) (percent) during the first 24 h and up to Day 7.
  Fraction of inspired oxygen (FiO2 [percent]). Results are shown as change from baseline, summarized at post-treatment time points.
  Definitions:
  FiO2=Fraction of inspired oxygen (percent); Baseline=The last pre-dose measurement taken on Day -1;
Time Frame: Post-treatment Day 1: 30 min, at 1h, 3h, 6h, 12h, 18h, 24 h; Day 2, 3, 5, and 7
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Fraction of inspired oxygen (percent)
Arm/Group | CHF5633 | Poractant Alfa
Number analyzed (Participants) | 56 | 57
Fraction of inspired oxygen (percent)
  Day 1, 30 min | 32.15 [27.91 to 36.39] | 34.08 [29.88 to 38.29]
  Day 1, 1 h | 31.41 [28.14 to 34.68] | 28.96 [25.76 to 32.16]
  Day 1, 3 h | 29.29 [26.05 to 32.52] | 28.87 [25.68 to 32.06]
  Day 1, 6 h | 27.76 [24.43 to 31.08] | 28.16 [24.88 to 31.45]
  Day 1, 12 h | 25.28 [22.71 to 27.85] | 28.05 [25.53 to 30.58]
  Day 1, 18 h | 26.18 [24.02 to 28.34] | 28.10 [25.97 to 30.23]
  Day 1, 24 h | 28.49 [25.02 to 31.96] | 29.50 [26.05 to 32.95]
  Day 2: number analyzed (Participants) | 56 | 55
  Day 2 | 29.29 [26.52 to 32.06] | 29.20 [26.46 to 31.93]
  Day 3: number analyzed (Participants) | 54 | 55
  Day 3 | 27.54 [23.64 to 31.44] | 29.07 [25.28 to 32.86]
  Day 5: number analyzed (Participants) | 54 | 52
  Day 5 | 28.06 [24.13 to 31.99] | 26.32 [22.41 to 30.23]
  Day 7: number analyzed (Participants) | 53 | 52
  Day 7 | 29.25 [25.22 to 33.28] | 28.02 [24.02 to 32.01]
Statistical Analysis 1: Comparison: CHF5633 vs Poractant Alfa; Day 1, 30 min post dose; Test type: Superiority; p = 0.519, Mixed model for repeated measurements; Mean Difference (Final Values) = -1.94, 95% CI 2-sided [-7.87 to 3.99]
Statistical Analysis 2: Comparison: CHF5633 vs Poractant Alfa; Day 1, 1 h post dose; Test type: Superiority; p = 0.282, Mixed model for repeated measurements; Mean Difference (Final Values) = 2.45, 95% CI 2-sided [-2.04 to 6.93]
Statistical Analysis 3: Comparison: CHF5633 vs Poractant Alfa; Day 1, 3 h post dose; Test type: Superiority; p = 0.854, Mixed model for repeated measurements; Mean Difference (Final Values) = 0.41, 95% CI 2-sided [-4.04 to 4.86]
Statistical Analysis 4: Comparison: CHF5633 vs Poractant Alfa; Day 1, 6 h post dose; Test type: Superiority; p = 0.861, Mixed model for repeated measurements; Mean Difference (Final Values) = -0.41, 95% CI 2-sided [-5.00 to 4.19]
Statistical Analysis 5: Comparison: CHF5633 vs Poractant Alfa; Day 1, 12 h post dose; Test type: Superiority; p = 0.117, Mixed model for repeated measurements; Mean Difference (Final Values) = -2.77, 95% CI 2-sided [-6.24 to 0.70]
Statistical Analysis 6: Comparison: CHF5633 vs Poractant Alfa; Day 1, 18 h post dose; Test type: Superiority; p = 0.185, Mixed model for repeated measurements; Mean Difference (Final Values) = -1.92, 95% CI 2-sided [-4.79 to 0.94]
Statistical Analysis 7: Comparison: CHF5633 vs Poractant Alfa; Day 1, 24 h post dose; Test type: Superiority; p = 0.678, Mixed model for repeated measurements; Mean Difference (Final Values) = -1.01, 95% CI 2-sided [-5.82 to 3.80]
Statistical Analysis 8: Comparison: CHF5633 vs Poractant Alfa; [analysis description as in outcome 1, analysis 8]; Test type: Superiority; p = 0.961, Mixed Models Analysis; Mean Difference (Final Values) = 0.09, 95% CI 2-sided [-3.49 to 3.67]
Statistical Analysis 9: Comparison: CHF5633 vs Poractant Alfa; Day 3, post dose; Test type: Superiority; p = 0.544, Mixed Models Analysis; Mean Difference (Final Values) = -1.53, 95% CI 2-sided [-6.53 to 3.46]
Statistical Analysis 10: Comparison: CHF5633 vs Poractant Alfa; Day 5, post dose; Test type: Superiority; p = 0.492, Mixed Models Analysis; Mean Difference (Final Values) = 1.74, 95% CI 2-sided [-3.28 to 6.76]
Statistical Analysis 11: Comparison: CHF5633 vs Poractant Alfa; Day 7, post dose; Test type: Superiority; p = 0.634, Mixed Models Analysis; Mean Difference (Final Values) = 1.23, 95% CI 2-sided [-3.90 to 6.36]

3. Primary Outcome: Number of Patients With Bronchopulmonary Dysplasia and Mortality
Description: Bronchopulmonary dysplasia and mortality.
  Results summarize the following items:
  Number of patients who died and the number of patients who had bronchopulmonary dysplasia (BPD) were assessed by treatment, at 36 weeks post menstrual age (PMA).
  Number of patients who died by Day 28 post-natal age (PNA).
  Number of patients with respiratory distress syndrome (RDS)-associated mortality by Day 14 post-natal age (PNA).
  Definitions:
  BPD=Bronchopulmonary dysplasia; Mortality/BPD incidence=The incidence of neonates dead within 36-week PMA or alive at 36-week PMA with a diagnosis of BPD; PMA=Post menstrual age; PNA=Post-natal age; RDS=Respiratory distress syndrome;
Time Frame: 36 weeks post menstrual age, Day 14 Post-Natal Age, Day 28 Post-Natal Age
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CHF5633 | Poractant Alfa
Number analyzed (Participants) | 56 | 57
Participants
  36 week PMA Incidence of BPD (Yes) | 31 | 32
  36 week PMA Mortality/BPD | 35 | 38
  36 week PMA Mortality | 4 | 6
  Day 28 (PNA) Mortality | 4 | 3
  Day 14 (PNA) RDS-associated mortality | 1 | 2
Statistical Analysis 1: Comparison: CHF5633 vs Poractant Alfa; Week 36 PMA Incidence of BPD; Test type: Superiority — Mortality or BPD incidence at 36-week PMA was compared by treatment, using Cochran-Mantel-Haenszel (CMH), adjusting for stratification gestational age (GA) group. Relative risk (RR) and its 95% confidence interval are also provided; p = 0.811, Cochran-Mantel-Haenszel; Relative risk = 1.03, 95% CI 2-sided [0.81 to 1.32]
Statistical Analysis 2: Comparison: CHF5633 vs Poractant Alfa; Week 36 PMA Incidence of Mortality/BPD; Test type: Superiority; p = 0.972, Cochran-Mantel-Haenszel; Relative risk = 1.00, 95% CI 2-sided [0.81 to 1.25]
Statistical Analysis 3: Comparison: CHF5633 vs Poractant Alfa; Week 36 PMA Mortality; Test type: Superiority; p = 0.619, Cochran-Mantel-Haenszel; Relative risk = 0.74, 95% CI 2-sided [0.23 to 2.42]
Statistical Analysis 4: Comparison: CHF5633 vs Poractant Alfa; Day 28 PNA Mortality; Test type: Superiority; p = 0.602, Cochran-Mantel-Haenszel; Relative risk = 1.46, 95% CI 2-sided [0.35 to 6.09]
Statistical Analysis 5: Comparison: CHF5633 vs Poractant Alfa; Day 14 PNA RDS-associated mortality in 14 days of life; Test type: Superiority; p = 0.606, Cochran-Mantel-Haenszel; Relative risk = 0.56, 95% CI 2-sided [0.06 to 5.29]

4. Other Pre Specified Outcome: Number of Patients With Normal Breathing (Room Air) Within 24 Hours
Description: Normal breathing (room air) within 24 hours
  The number of patients with at least one reading of FiO2 equal to 21% (i.e. corresponding to room air for oxygen concentration) within 24 hours from first dose of surfactant was evaluated.
Time Frame: Post-treatment up to 24 h
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CHF5633 | Poractant Alfa
Number analyzed (Participants) | 56 | 57
Participants | 38 | 43
Statistical Analysis 1: Comparison: CHF5633 vs Poractant Alfa; Test type: Superiority; p = 0.409, Fisher Exact; Odds Ratio (OR) = 0.69, 95% CI 2-sided [0.30 to 1.57]

5. Other Pre Specified Outcome: Number of Patients With the Need for Re-dosing (Use of Rescue Surfactant)
Description: Number of patients with the need for re-dosing (use of rescue surfactant).
  The number of patients requiring at least one surfactant rescue dose (i.e. re-dosing with the study drug) at any time during the study was evaluated.
Time Frame: Day 1 to Day 7
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | CHF5633 | Poractant Alfa
Number analyzed (Participants) | 56 | 57
Participants
  Patients receiving rescue at any time during the study | 19 | 17
  1 rescue dose given | 11 | 12
  2 rescue doses given | 8 | 5
Statistical Analysis 1: Comparison: CHF5633 vs Poractant Alfa; The percentage of patients requiring at least one rescue surfactant dose; Test type: Superiority — The percentage of patients requiring at least one rescue surfactant dose were compared by treatment group using the Fisher's exact test at 5% significance interval. Odds ratio (OR) and related exact 95% CI are also provided; p = 0.689, Fisher Exact; Odds Ratio (OR) = 1.21, 95% CI 2-sided [0.55 to 2.67]

6. Other Pre Specified Outcome: Time to Reach Normal Breathing (Room Air) Within 24 Hours
Description: Time to reach normal breathing (room air) within 24 hours.
  The median time to reach normal breathing (room air) within 24 hours from first dose of surfactant was evaluated. These are the patients who contributed to the results in the outcome measure 'Normal Breathing (room air) within 24 hours'.
Time Frame: Post-treatment Day 1: up to 24 h
Population: as for outcome 1
Measure: Median (Full Range); unit: hour
Arm/Group | CHF5633 | Poractant Alfa
Number analyzed (Participants) | 38 | 43
hour | 2.980 [0.38 to 24.00] | 2.320 [0.22 to 24.00]
Statistical Analysis 1: Comparison: CHF5633 vs Poractant Alfa; Test type: Superiority; p = 0.935, Wilcoxon (Mann-Whitney)

7. Other Pre Specified Outcome: Concentration of Biomarkers of Inflammation in Tracheal Aspirates
Description: The inflammatory status of the patients was assessed (in a subgroup of babies who required endotracheal intubation for mechanical ventilation, when feasible). This was performed by measuring the concentration of specific biomarkers of inflammation in tracheal aspirates. The biomarkers measured were: Interleukin 1β, Interleukin 6, Interleukin 8, Myeloperoxidase, and Tumor Necrosis Factor-Alpha.
  The total protein content in tracheal aspirates was measured as an endogenous marker of dilution to calculate the extent to which epithelial lining fluid (ELF) was diluted during the tracheal aspirate procedure. To adjust for variation during the collection of tracheal aspirates, the measured cytokines values were normalized to the total protein. Results are presented as change from baseline in pg/mg total protein and were evaluated by descriptive statistics.
  Definition:
  Baseline=The last pre-dose measurement taken on Day -1;
Time Frame: Post-treatment Day 1 (24 h), Day 2 (48 h)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: pg/mg total protein
Arm/Group | CHF5633 | Poractant Alfa
Number analyzed (Participants) | 56 | 57
pg/mg total protein
  Interleukin 1β, Day 1, 24 h: number analyzed (Participants) | 14 | 12
  Interleukin 1β, Day 1, 24 h | -38.535 (93.111) | -39.896 (134.659)
  Interleukin 1β, Day 2, 48 h: number analyzed (Participants) | 13 | 9
  Interleukin 1β, Day 2, 48 h | 3.681 (154.736) | -40.564 (158.194)
  Interleukin 6, Day 1, 24 h: number analyzed (Participants) | 14 | 13
  Interleukin 6, Day 1, 24 h | -200.074 (761.436) | -792.196 (2657.394)
  Interleukin 6, Day 2, 48 h: number analyzed (Participants) | 13 | 9
  Interleukin 6, Day 2, 48 h | -129.368 (954.282) | -1089.753 (3222.013)
  Interleukin 8, Day 1, 24 h: number analyzed (Participants) | 14 | 13
  Interleukin 8, Day 1, 24 h | 389.86 (5240.76) | -843.74 (4720.36)
  Interleukin 8,Day 2, 48 h: number analyzed (Participants) | 13 | 9
  Interleukin 8,Day 2, 48 h | 821.16 (5978.87) | -243.71 (6425.90)
  Myeloperoxidase, Day 1, 24 h: number analyzed (Participants) | 11 | 10
  Myeloperoxidase, Day 1, 24 h | 267337.7 (399695.4) | 52663.5 (264660.9)
  Myeloperoxidase, Day 2, 48 h: number analyzed (Participants) | 10 | 8
  Myeloperoxidase, Day 2, 48 h | 310323.0 (419874.0) | 508378.1 (381999.8)
  Tumor Necrosis Factor-Alpha, Day 1, 24 h: number analyzed (Participants) | 13 | 12
  Tumor Necrosis Factor-Alpha, Day 1, 24 h | -16.047 (42.924) | -19.985 (67.539)
  Tumor Necrosis Factor-Alpha, Day 2, 48 h: number analyzed (Participants) | 11 | 9
  Tumor Necrosis Factor-Alpha, Day 2, 48 h | 2.899 (71.215) | -25.573 (78.934)

8. Other Pre Specified Outcome: Immunogenicity: Assessment of Antibodies to Surfactant Protein B (SP-B) Analogue (CHF 5736.03) and to Surfactant Protein C (SP-C) Analogue (CHF 4902.03)
Description: Immunogenicity was assessed by measuring antibodies to SP-B analogue (CHF 5736.03) and to SP-C analogue (CHF 4902.03), contained in CHF 5633.
  Results are expressed as the titre (i.e. serum dilution) at which the sample had an absorbance of 0.069 (background) for SP-C Analogue (CHF 4902.03) CHF or an absorbance of 0.05 for SP-B Analogue (CHF 5736.03) in a microplate reader. The positive control serum was diluted in buffer solution and the maximum binding for the positive control was determined at dilutions < 1/12.5 for SPC and <1/100 for SPB. Test samples for immunogenicity were analyzed by using negative and positive controls. By definition, titer <12.5 for CHF-4902.03 and <100 for CHF-5736.02 show that the test serum had an absorbance equal to background at the same dilution at which the positive control had the maximum binding, implying absence of antibodies.
Time Frame: At approximately 5 weeks after the administration of study drug (with a range from 3 to 6 weeks).
Population: Safety Population. All randomized patients who took at least one dose of study medication and who had the assessment done on 28 day PNA.
Measure: Number; unit: Titre (dilution with 0.050 absorbance)
Arm/Group | CHF5633 | Poractant Alfa
Number analyzed (Participants) | 60 | 61
Titre (dilution with 0.050 absorbance)
  Antibody to SP-B (CHF 5736.03): number analyzed (Participants) | 53 | 54
  Antibody to SP-B (CHF 5736.03) | 100 | 100
  Antibody to SP-C (CHF 4902.03): number analyzed (Participants) | 53 | 54
  Antibody to SP-C (CHF 4902.03) | 12.5 | 12.5

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the time of the informed consent signature* up to the study completion or discontinuation. The study duration was from minutes after birth and up to 36 week post menstrual age (PMA) *The written informed consent was obtained from parents/legal representative (according to local regulation) prior to any study-related procedures.
Description: Analysis of adverse events (AEs) was performed on treatment emergent AEs (TEAEs).
  Safety population=All randomized subjects who received at least one dose of study treatment, was used for the evaluation of adverse events.
  An Independent Safety Monitoring Board (ISMB) was established on an ongoing basis to ensure the safety of study patients, with regard to the incidence of major adverse outcomes after the administration of the study drug (such as serious adverse events [SAEs]).
Arm/Group | CHF5633 | Poractant Alfa
All-Cause Mortality (participants affected / at risk) | 4/59 | 7/58
Serious Adverse Events (participants affected / at risk) | 20/59 | 20/58
Other Adverse Events (participants affected / at risk) | 59/59 | 58/58
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHF5633 (N=59) | Poractant Alfa (N=58)
Disseminated intravascular coagulation in newborn (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Bradycardia neonatal (Cardiac disorders) | 1 (1) | 0 (0)
Amniotic band syndrome (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Cerebellar hypoplasia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Congenital cytomegalovirus infection (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Developmental glaucoma (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Retinopathy of prematurity (Eye disorders) | 2 (2) | 1 (1)
Neonatal intestinal perforation (Gastrointestinal disorders) | 2 (2) | 3 (3)
Necrotising enterocolitis neonatal (Gastrointestinal disorders) | 1 (1) | 3 (3)
Neonatal gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pneumoperitoneum (Gastrointestinal disorders) | 0 (0) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Neonatal pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Respiratory syncytial virus infection (Infections and infestations) | 0 (0) | 1 (1)
Serratia bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Sepsis neonatal (Infections and infestations) | 4 (5) | 2 (2)
Urinary tract infection neonatal (Infections and infestations) | 1 (2) | 0
Feeding disorder neonatal (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 1 (1) | 3 (3)
Cerebral haemorrhage neonatal (Nervous system disorders) | 1 (1) | 2 (2)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Oliguria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal failure neonatal (Renal and urinary disorders) | 1 (1) | 0 (0)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Atelectasis neonatal (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Tracheal stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Neonatal hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CHF5633 (N=59) | Poractant Alfa (N=58)
Anaemia neonatal (Blood and lymphatic system disorders) | 49 (52) | 47 (50)
Bandaemia (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Leukocytosis (Blood and lymphatic system disorders) | 4 (5) | 7 (7)
Neutropenia neonatal (Blood and lymphatic system disorders) | 2 (2) | 4 (4)
Thrombocytopenia neonatal (Blood and lymphatic system disorders) | 16 (18) | 16 (17)
Thrombocytosis (Blood and lymphatic system disorders) | 2 (2) | 3 (3)
Bradycardia neonatal (Cardiac disorders) | 11 (11) | 8 (8)
Neonatal tachycardia (Cardiac disorders) | 3 (3) | 5 (5)
Tricuspid valve incompetence (Cardiac disorders) | 3 (3) | 3 (3)
Adrenal insufficiency neonatal (Congenital, familial and genetic disorders) | 4 (5) | 3 (3)
Atrial septal defect (Congenital, familial and genetic disorders) | 21 (22) | 19 (21)
Hydrocele (Congenital, familial and genetic disorders) | 4 (4) | 1 (1)
Patent ductus arteriosus (Congenital, familial and genetic disorders) | 26 (26) | 34 (37)
Sickle cell trait (Congenital, familial and genetic disorders) | 4 (4) | 0 (0)
Hypothyroidism (Endocrine disorders) | 2 (2) | 5 (5)
Transient hypothyroxinaemia of prematurity (Endocrine disorders) | 2 (2) | 3 (3)
Retinopathy of prematurity (Eye disorders) | 20 (24) | 18 (18)
Abdominal distension (Gastrointestinal disorders) | 7 (7) | 5 (5)
Constipation (Gastrointestinal disorders) | 5 (5) | 5 (5)
Gastrointestinal hypomotility (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrointestinal motility disorder (Gastrointestinal disorders) | 3 (3) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 8 (8) | 5 (5)
Haematochezia (Gastrointestinal disorders) | 4 (4) | 3 (3)
Inguinal hernia (Gastrointestinal disorders) | 9 (9) | 9 (9)
Umbilical hernia (Gastrointestinal disorders) | 3 (3) | 2 (2)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 4 (4)
Vomiting (Gastrointestinal disorders) | 2 (2) | 3 (3)
Peripheral oedema neonatal (General disorders) | 4 (4) | 5 (5)
Hyperbilirubinaemia neonatal (Hepatobiliary disorders) | 40 (44) | 32 (35)
Jaundice cholestatic (Hepatobiliary disorders) | 0 (0) | 3 (3)
Bacterial disease carrier (Infections and infestations) | 1 (1) | 3 (3)
Neonatal pneumonia (Infections and infestations) | 7 (8) | 5 (7)
Oral candidiasis (Infections and infestations) | 3 (5) | 1 (1)
Sepsis neonatal (Infections and infestations) | 13 (14) | 17 (23)
Staphylococcal bacteraemia (Infections and infestations) | 3 (3) | 1 (1)
Tracheitis (Infections and infestations) | 1 (2) | 3 (3)
Urinary tract infection neonatal (Infections and infestations) | 5 (5) | 8 (9)
Skin abrasion (Injury, poisoning and procedural complications) | 3 (3) | 2 (3)
Blood creatinine increased (Investigations) | 3 (3) | 2 (2)
Blood urea increased (Investigations) | 3 (3) | 1 (1)
C-reactive protein increased (Investigations) | 4 (5) | 7 (10)
Chest X-ray abnormal (Investigations) | 6 (6) | 1 (1)
Alkalosis hypochloraemic (Metabolism and nutrition disorders) | 1 (1) | 3 (3)
Feeding disorder neonatal (Metabolism and nutrition disorders) | 5 (5) | 3 (3)
Feeding disorder of infancy or early childhood (Metabolism and nutrition disorders) | 2 (3) | 3 (3)
Hypercalcaemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 20 (26) | 13 (16)
Hyperkalaemia (Metabolism and nutrition disorders) | 5 (6) | 8 (9)
Hypermagnesaemia (Metabolism and nutrition disorders) | 4 (4) | 7 (7)
Hypernatraemia (Metabolism and nutrition disorders) | 16 (20) | 10 (10)
Hypocalcaemia (Metabolism and nutrition disorders) | 9 (11) | 9 (10)
Hypoglycaemia neonatal (Investigations) | 8 (8) | 10 (12)
Hypokalaemia (Metabolism and nutrition disorders) | 12 (14) | 7 (7)
Hypophosphataemia (Metabolism and nutrition disorders) | 5 (5) | 5 (5)
Metabolic acidosis (Metabolism and nutrition disorders) | 18 (19) | 23 (23)
Metabolic alkalosis (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Neonatal hyponatraemia (Metabolism and nutrition disorders) | 17 (23) | 19 (21)
Poor feeding infant (Metabolism and nutrition disorders) | 2 (2) | 6 (6)
Osteopenia (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 3 (3)
Cerebral ventricle dilatation (Nervous system disorders) | 3 (3) | 3 (3)
Convulsion neonatal (Nervous system disorders) | 6 (7) | 5 (5)
Intraventricular haemorrhage neonatal (Nervous system disorders) | 18 (22) | 19 (23)
Jaundice neonatal (Pregnancy, puerperium and perinatal conditions) | 9 (9) | 14 (16)
Leukopenia neonatal (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 4 (4)
Agitation neonatal (Psychiatric disorders) | 7 (7) | 3 (3)
Hydronephrosis (Renal and urinary disorders) | 4 (4) | 3 (3)
Apnoea neonatal (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 13 (13)
Atelectasis neonatal (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 5 (5)
Bronchopulmonary dysplasia (Respiratory, thoracic and mediastinal disorders) | 33 (35) | 32 (32)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 3 (4) | 2 (2)
Neonatal hypoxia (Respiratory, thoracic and mediastinal disorders) | 11 (11) | 11 (12)
Neonatal respiratory acidosis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 7 (8)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 13 (14) | 12 (13)
Neonatal respiratory failure (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 6 (6)
Neonatal tachypnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Pulmonary interstitial emphysema syndrome (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 4 (4)
Pulmonary oedema neonatal (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2)
Dermatitis diaper (Skin and subcutaneous tissue disorders) | 5 (7) | 8 (10)
Hypertension neonatal (Vascular disorders) | 3 (3) | 3 (3)
Neonatal hypotension (Vascular disorders) | 18 (22) | 17 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Chiesi Farmaceutici S.p.A. (Sponsor) can publish or present results of this study at scientific meetings and submit the data to national and international Regulatory Authorities. The Sponsor reserves the right to use the data for industry purposes. Investigators will inform the Sponsor before using the results of the study for publication or presentation, and will provide the Sponsor with a copy of the proposed presentation. Data from individual study sites must not be published separately.

DOCUMENTS (2):
  • Study Protocol (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/76/NCT02452476/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-18): https://cdn.clinicaltrials.gov/large-docs/76/NCT02452476/SAP_001.pdf